CLINICAL TRIAL: NCT05444426
Title: Investigation of the Effect of Conventional Treatment on Postural Stability and Balance in Individuals With Shoulder Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Medipol University (Other)
Responsible Party: Principal Investigator, Tuğçe Tahmaz, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Shoulder Pain
Record Dates: First submitted 2022-06-30; First posted 2022-07-05 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Shoulder Pain; Balance; Distorted
Keywords: shoulder pain; balance; postural stability
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): A 24-session physiotherapy program will be applied to the patients in the treatment group.
  The conventional physiotherapy program of the patients in the treatment group; will consist of 20 minutes of the hot pack, 20 minutes of conventional TENS (COMPEX Rehab 400), 1 MHz frequency, 1.5 W/cm² intensity ultrasound (Chattanooga Intelect Ultrasound) on the shoulder joint for 5 minutes. In the exercise program; A combined exercise program including active assistive and active range of motion exercises, stretching exercises for the shoulder muscles at the pain limit and posture exercises will be applied. As the severity of pain decreases, strengthening exercises for the rotator cuff and scapulary muscles will be given.
  Interventions: Other: Shoulder Rehabilitation
- Control Group (No Intervention): Pain, Active range of motion, balance, and postural stability will be assessed in the first week .

INTERVENTIONS:
Other: Shoulder Rehabilitation — hot pack, conventional TENS (COMPEX Rehab 400), 1 MHz frequency, 1.5 W/cm² intensity ultrasound (Chattanooga Intelect Ultrasound), active assistive and active range of motion exercises, stretching exercises for the shoulder muscles at the pain limit and posture exercises will be applied.
  Arms: Treatment Group

SUMMARY:
Shoulder pain is one of the most common musculoskeletal complaints that people need treatment for. Typical signs and symptoms include pain during reaching, muscle weakness, and interrupted sleep. The shoulder is one of the most common areas of pain, ranking third among musculoskeletal pains in the general population. There is a lack of information regarding the impact of shoulder-related problems on the general population, and therefore there is a growing interest in identifying adverse factors associated with shoulder problems. In our study, the postural stability and balance status of individuals with shoulder pain complaints will be evaluated and the effects of conventional treatment of shoulder pain on postural instability and balance parameters will be investigated.

DETAILED DESCRIPTION:
The muscle that is important in lateral flexion of the trunk is the latissimus dorsi. There is a hypothesis that this muscle acts as a force transmitter from the gluteus maximus muscle to the upper extremity via myofascial connections. In the study of Kaur et al., it was reported that the myofascial connection between the hip muscles and the lateral flexors of the trunk increases the serratus anterior muscle activation. Therefore, deterioration in the performance of trunk muscles may affect the activation of the serratus anterior, resulting in decreased scapular upward rotation and posterior tilt, which may contribute to the development of pain and shoulder injury. Decreased core endurance can result in poor transmission of force generated in the lower body to the upper body and may contribute to upper limb incorrect positioning. 40 individuals with shoulder pain symptoms were planned to participate in the study. The individuals included in the study were divided into two groups the treatment group and the control group. A 24-session physiotherapy program will be applied to the patients in the treatment group. Pain, active joint range of motion, balance, and postural stability will be evaluated first week and eighth weeks.

ELIGIBILITY:
Inclusion Criteria:

* Having a complaint of shoulder pain for at least 3 months
* Being between the ages of 19-60

Exclusion Criteria:

* Having had a surgical operation in the last 6 months,
* Having cognitive problems that prevent participation in exercises.

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Change of postural stability from baseline to 8 weeks | 8 weeks
  Biodex Balance system will be used to evaluate the postural stability and balance of individuals.
  In evaluating the Biodex Balance System, the postural stability test of the participants will be assessed on the dynamic platforms. In the fall risk assessment, it will be evaluated with eyes open and eyes closed on the dynamic platform, which increases its mobility from 12th to 6th Levels. During the test, participants will be asked to look at a fixed point at eye level. The test will be repeated 3 times and the average will be taken. A 15-second rest period will be given between each repetition.

SECONDARY OUTCOMES:
Change of Pain Level from baseline to 8 weeks | 8 weeks
  A 'Numerical Analog Scale' will be used in the assessment of pain. The Numeric Pain Rating Scale (NPRS) (an outcome measure) that is a unidimensional measure of pain intensity in adults, including those with chronic pain due to rheumatic diseases. The NPRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain.The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
Change of shoulder joint range baseline to 8 weeks | 8 weeks
  A universal goniometer will be used in the assessment of active joint range of motion.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rosa DP, Borstad JD, Ferreira JK, Gava V, Santos RV, Camargo PR. Comparison of specific and non-specific treatment approaches for individuals with posterior capsule tightness and shoulder impingement symptoms: A randomized controlled trial. Braz J Phys Ther. 2021 Sep-Oct;25(5):648-658. doi: 10.1016/j.bjpt.2021.04.003. Epub 2021 May 4. PMID 34001426
- [Background] Ostor AJ, Richards CA, Prevost AT, Speed CA, Hazleman BL. Diagnosis and relation to general health of shoulder disorders presenting to primary care. Rheumatology (Oxford). 2005 Jun;44(6):800-5. doi: 10.1093/rheumatology/keh598. Epub 2005 Mar 15. PMID 15769790
- [Background] Carvalhais VO, Ocarino Jde M, Araujo VL, Souza TR, Silva PL, Fonseca ST. Myofascial force transmission between the latissimus dorsi and gluteus maximus muscles: an in vivo experiment. J Biomech. 2013 Mar 15;46(5):1003-7. doi: 10.1016/j.jbiomech.2012.11.044. Epub 2013 Feb 8. PMID 23394717
- [Background] Kaur N, Bhanot K, Brody LT, Bridges J, Berry DC, Ode JJ. Effects of lower extremity and trunk muscles recruitment on serratus anterior muscle activation in healthy male adults. Int J Sports Phys Ther. 2014 Dec;9(7):924-37. PMID 25540708